CLINICAL TRIAL: NCT05234905
Title: Oncolytic Virus(H101) Combined With Camrelizumab for Recurrent Cervical Cancer: a Prospective, Multicenter Study
Brief Title: H101 Combined With Camrelizumab for Recurrent Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARTOnG 2105
Record Dates: First submitted 2022-01-27; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-12

CONDITIONS: Uterine Cervical Neoplasms; Oncolytic Virotherapy; Camrelizumab
Keywords: Recurrent cervical cancer; H101; Camrelizumab; Objective response rate
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant human adenovirus type 5+ Camrelizumab (Experimental): Recombinant human adenovirus type 5: one lesion was selected for intratumoral injection.Intratumoral injection of H101 was performed on day 1 and day 4 of each cycle, and was repeated once every 3 weeks. H101 dose:
  ① Tumor maximum diameter ≤5cm, 1.5×10^12vp (3 injections) on day 1, 1.0×10^12vp (2 injections) on day 4.
  ② Tumor maximum diameter >5cm but ≤10cm, 3.0×10^12vp (6 injections) on day 1 and 2.0×10^12vp (4 injections) on day 4.
  ③ Tumor maximum diameter >10cm, 4.5×10^12vp (9 injections) on day 1 and 3.0×10^12vp (6 injections) on day 4.
  H101 intratumoral injection until the tumor is completely regressed to stop the drug, but not more than 5 cycles at most.
  Camrelizumab: administered after H101 on day 1 of each cycle and repeated for 3 weeks. Camrelizumab dose: 200 mg IV.
  Interventions: Drug: Recombinant human adenovirus type 5＋Camrelizumab

INTERVENTIONS:
Drug: Recombinant human adenovirus type 5＋Camrelizumab — Recombinant human adenovirus type 5: one lesion was selected for intratumoral injection.Intratumoral injection of H101 was performed on day 1 and day 4 of each cycle, and was repeated once every 3 weeks. H101 dose:
  ① Tumor maximum diameter ≤5cm, 1.5×1012vp (3 injections) on day 1, 1.0×1012vp (2 injections) on day 4.
  ② Tumor maximum diameter >5cm but ≤10cm, 3.0×1012vp (6 injections) on day 1 and 2.0×1012vp (4 injections) on day 4.
  ③ Tumor maximum diameter >10cm, 4.5×1012vp (9 injections) on day 1 and 3.0×1012vp (6 injections) on day 4.
  H101 intratumoral injection until the tumor is completely regressed to stop the drug, but not more than 5 cycles at most.
  Camrelizumab: administered after H101 on day 1 of each cycle and repeated for 3 weeks. Camrelizumab dose: 200 mg IV.
  Other Names: H101＋Camrelizumab

SUMMARY:
There is no standard treatment for recurrent cervical cancer that progresses or persists after first-line treatment. The objective response rate of anti-PD-1 antibody treatment is about 15%. The purpose of this study was to evaluate whether the regimen could improve the objective response rate by intratumoral injection of oncolytic virus(recombinant human adenovirus type 5 injection, H101) combined with anti-PD-1 antibody(camrelizumab).

DETAILED DESCRIPTION:
1. Main research purpose To evaluate the efficacy of H101 combined with camrelizumab in patients with incurable recurrent cervical cancer.
2. Secondary research purpose To evaluate other curative effects of H101 combined with camrelizumab in patients with incurable recurrent cervical cancer.

   To evaluate the safety of H101 combined with camrelizumab in patients with incurable recurrent cervical cancer.
3. Purpose of Exploratory Research To explore the changes of tumor microenvironment before and after H101 injection and the mechanism of action in combination with PD-1, and to accurately screen the beneficiaries based on molecular expression.
4. Overall experimental design This study is a multicenter, prospective, clinical study to investigate the efficacy and safety of H101 combined with camrelizumab in the treatment of incurable recurrent cervical cancer patients. It is expected that 55 subjects will be enrolled.

   The study was divided into 5 phases: screening period, baseline period, treatment period, and follow-up period. Patients with recurrent cervical cancer who were eligible for inclusion and were incurable by previous first-line treatment were screened. During the follow-up period, follow-up was conducted every 1 month for at least 2 years.
5. Subject population The target population of this study was patients with recurrent cervical squamous cell carcinoma/adenocarcinoma/adenosquamous carcinoma who were incurable after first-line therapy.
6. Treatment allocation All subjects enrolled in this study received H101 combined with camrelizumab.
7. Drug dosage and administration in the trial Dosing regimen: H101 + camrelizumab. 1) H101: 1 lesion was selected for intratumoral injection. Intratumoral injection of H101 was used on the 1st and 4th day of each cycle, repeated once in 3 weeks. H101 dosage: Tumor maximum diameter ≤5 cm, 1.5×10^12vp (3 injections) on day 1 and 1.0×10^12vp (2 injections) on day 4.

Tumor maximum diameter >5cm but ≤10cm, 3.0×10^12vp (6 injections) on day 1, 2.0×10^12vp (4 injections) on day 4.

Tumor maximum diameter >10cm, 4.5×10^12vp (9 injections) on day 1 and 3.0×10^12vp (6 injections) on day 4.

H101 will be used until injected lesion disappears or 5 cycles, whichever occurs first.

2) Camrelizumab: 200 mg intravenously. Dosing after H101 on day 1 of each cycle, repeated 3 weeks. The drug was discontinued or discontinued for 2 years until the patient developed tumor progression or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met for inclusion:

1. Participants voluntarily participated in this study and signed the informed consent;
2. 18-80 years old;
3. Cervical squamous cell carcinoma/adenocarcinoma/adenosquamous carcinoma;
4. Participants with incurable recurrence after first-line treatment or participants with incurable recurrence within the irradiation field;
5. At least one lesion that meets RICIST 1.1 criteria can be evaluated and can be injected intratumorally;
6. ECOG score 0-2 points;
7. Expected survival > 3 months;
8. Women of childbearing age must undergo a pregnancy test (serum or urine) before enrollment, and the result is negative, and they are willing to use appropriate methods of contraception during the trial;
9. Those who can tolerate and comply with the trial protocol, as determined by the investigator.

Exclusion Criteria:

Those who have one of the following conditions should be excluded and cannot be selected:

1. There is an infection at the intended injection site;
2. Liver cirrhosis, decompensated liver disease;
3. Have a history of immunodeficiency, including HIV positive or other acquired congenital immunodeficiency diseases;
4. Chronic renal insufficiency and renal failure;
5. Combined with other malignant tumor patients who still need treatment and/or newly diagnosed within 5 years;
6. Myocardial infarction, severe arrhythmia and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification);
7. Complications, need to take drugs with serious liver and kidney damage during treatment, such as tuberculosis;
8. Previous use of anti-PD-1 drugs or oncolytic viruses;
9. Patients who cannot understand the experimental content and cannot cooperate and those who refuse to sign the informed consent;
10. Those with concomitant diseases or other special conditions that seriously endanger the safety of patients or affect the completion of the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective Response Rate) | 2 years
  The proportion of CR(complete response) and PR(partial response) in all patients.

SECONDARY OUTCOMES:
PFS(Progression Free Survival) | 2 years
  Refers to the time from the first treatment day to the first occurrence of disease progression or death from any cause (whichever occurs first), and the end point event is determined by the investigator according to RECIST v1.1.
DCR(Disease Control Rate) | 2 years
  The proportion of CR(complete response), PR(partial response) and SD(stable disease) in all patients.
OS(Overall Survival) | 2 years
  Time between the date of randomization grouping and death from any cause or the end of the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Zhang, Study Director — Zhejiang Cancer Hospital
Locations (4):
- China (4):
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospital Medical Group, Jinhua
  - Ningbo First Hospital, Ningbo
  - Taizhou Central Hospiatl, Taizhou

IPD SHARING:
Plan to Share IPD: No